CLINICAL TRIAL: NCT01548963
Title: Perioperative Versus Postoperative Glycemia Control in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Blaha, MD, PhD., Principal Investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: eMPC_long
Record Dates: First submitted 2012-02-25; First posted 2012-03-08 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Perioperative and Postoperative Hyperglycemia; Tight Glycemia Control
Keywords: Tight glycemia control; Model Predictive Control algorithm; Cardiac surgery patients
MeSH Terms: interventions — Glycemic Control

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perioperative glycemia control (Experimental): Group of perioperative intensive glycemia control: blood glucose level will be maintained by continuous insulin infusion (Actrapid, Novo Nordisk A/S, Bagsvaerd, Danemark - 50 IU/50 ml FR) according to actual glycemia to keep it within normoglycemia limits (4.4 - 6.1 mmol/l) since patient's admission to operating room. Samplings will be taken in 1 to 4 hours intervals in accordance with glycemia stability and MPC algorithm suggestions.
  Interventions: Procedure: Intensive glycemia control
- Postoperative glycemia control (Active Comparator): Group of standard glycemia control: blood glucose level will be maintained by continuous insulin infusion (see above) within normoglycemia limits (4.4 - 6.1 mmol/l) after patient's admission to ICU after cardiac surgery. During surgery hyperglycemia will not be interfered before it will reach level of 10 mmol/l.
  Interventions: Procedure: Intensive glycemia control

INTERVENTIONS:
Procedure: Intensive glycemia control — Blood glucose levels will be maintained by continuous insulin infusion (Actrapid, Novo Nordisk A/S, Bagsvaerd, Danemark - 50 IU/50 ml FR) within normoglycemia limits (4.4 - 6.1 mmol/l)
  Other Names: Tight glycemia control; Blood glucose control

SUMMARY:
It is known that acute stress of organism often leads to hyperglycemia even in nondiabetic patients. It is also known that pathophysiological mechanisms: enhanced gluconeogenesis, impaired insulin secretion and decreased insulin sensitivity due to anti-insulin effect of stress hormones and proinflammatory cytokines, or changes of glucose excretion and renal tubular resorption.

Many studies proved the negative effects of hyperglycemia to different tissues and organs, e.g. hearth (increasing size of myocardial necrosis, reducing coronary collateral blood flow, exaggerating ischemia-reperfusion injury, impairing ischemic preconditioning), vascular (increased risk of thrombosis, endothelial dysfunction, activation of systemic inflammation with destabilization of atherosclerotic plaques), kidneys and its association with infectious complications.

The first Leuven study (published in 2001) demonstrated that hyperglycemia in critical care patients significantly increases risk of organ complication and total mortality. Although the importance of postoperative tight glycemia control is now widely accepted, glycemia stability during cardiac surgery is often neglected. It is known that postoperative hyperglycemia has negative effects, but it is not known what effect has its peroperative elevation.

Goal of this study is to demonstrate, whether full perioperative intensive glycemia control can reduce the incidence of postoperative morbidity even more than postoperative glycemia control only.

DETAILED DESCRIPTION:
It has been for a long time a well known phenomenon that the acute stress of organism induced for instance by an extensive surgery often leads to hyperglycemia, even in patients without a previous history of diabetes. Also well known are the common pathophysiological mechanisms, which are responsible for this, such as enhanced hepatic gluconeogenesis, impaired insulin secretion and decreased insulin sensitivity due to anti-insulin effect of stress hormones and proinflammatory cytokines, or a change of glucose excretion and higher renal tubular resorption.

Many studies proved the negative effect of the elevated blood glucose level to different tissues and organs. Even short-term hyperglycemia has been found to markedly impair cardiovascular function in ischemic heart, increasing size of myocardial necrosis, reducing coronary collateral blood flow, exaggerating ischemia-reperfusion cellular injury and/or impairing ischemic preconditioning.

Also other studies have identified numerous hyperglycemia-induced abnormalities such as increased risk of thrombosis, endothelial disfunction or activation of systemic inflammation, with possible destabilization of atherosclerotic plaques leading to acute ischemic syndromes. Hyperglycemia also has effect to the extent of renal injury, e.g. in patients after cardiac surgery, and last but not least, hyperglycemia has been associated with increased postoperative infectious complications.

Despite all those facts hyperglycemia has been until recently considered as a "protective" mechanism for patients in critical condition, when the cells are offered a supranormal amount of easily accessible energy. This approach has been radically changed thanks to Leuven study published by prof.Van den Berghe and her colleagues in 2001 in New England Journal of Medicine. This fundamental study proved that a higher levels of blood glucose in intensive care patients significantly increase the risk of organ complications as well as an overall death rate, and that, on the contrary, we can significantly decrease both mortality, as well as the amount of organ complications connected with the critical state by an intensive insulin therapy aimed to keep normoglycemia. Such results were confirmed also by another study of prof.Van den Berghe and her colleagues (published in NEJM 2006), this time performed on non-surgery patients. This fact was quickly accepted by the intensivists and therefore it is nowadays commonplace for us to carefully monitor blood glucose levels in postoperative ICU, and keep it at normal levels.

Both the above-mentioned studies are even more significant for cardiac surgery patients, since the population of the patients in the first Leuven study (2001), where the results of intensive insulinotherapy were more distinct in comparison with non-surgery population (2006) mostly thanks to a 40% reduced mortality, consisted up to 63% from patients following cardiac surgery.

If normoglycemia is commonplace in postoperative intensive care, then the stability of glycemia during cardiac surgery is usually neglected. There is no clear recommendation regarding when it is suitable to start intensive control of glycemia, whether to do so after the surgery or already during the surgery. We know that postoperative hyperglycemia has many negative effects on the organism, however, we do not know yet whether the peroperative rise of blood glucose itself during cardiac or other extensive surgery with postoperative maintenance of normoglycemia has negative or benefiting effects on the organism. Until now, there has not yet been a valid study performed that would answer this concrete question.

THE GOALS OF THE PROJECT:

The goal of this study is to prove whether by full perioperative intensive control of glycemia, the occurrence of organ complications will be decreased even more significantly than by only postoperative normalization of hyperglycemia, what has already been proved by published studies. This proposed study is aiming at complementing the fundamental Leuven study with perioperative data and therefore answering the question, when to start the control of glycemia by an intensified insulinotherapy in patients undergoing cardiac surgery.

A decisive factor for the success of the project is also a quality protocol of glycemia control in perioperative care. During the previous years there were a number of various insulin protocols that more or less successfully tried to keep the levels of blood glucose in normoglycemia. Thanks to the European study of CLINICIP (Closed Loop Insulin Infusion for Critically Ill Patients) our Department took part in as a clinical partner, the investigators had the possibility to evaluate several European protocols and to compare them with the computer algorithm MPC (Model Predictive Control). The comparison of the possibilities to keep the levels of blood glucose in normoglycemia ended positively in favors of eMPC algorithm compare to the standard protocols. Therefore the investigators decided to use its adaptative version also in this project for glycemia control.

THE HYPOTHESIS AND EXPECTED RESULTS:

The investigators hypothesize, that if the postoperative normalization of already started hyperglycemia can significantly decreases the occurrence of postoperative complications, then absolute perioperative glycemia control, thanks to complete blockage of the negative influences of even the short term hyperglycemia, can even further emphasize the reduction of the postoperative complications.

OUTCOME MEASURES:

Primary outcome - to prove, whether the full blocking of the perioperative blood glucose elevation will reach a lower occurrence of postoperative organ complications, than in patients with a temporary peroperative rise of glycemia. The investigators will observe a number of adverse events (newly developed organ dysfunctions) from any cause during the postoperative hospital stay:

cardiovascular (LCO, postoperatively initiated inotropic support or intra-aortic balloon counterpulsation, acute myocardial ischemia, moderate to severe arrhythmias, cardiopulmonary resuscitation), respiratory (acute pneumonia, fluidothorax > 300 ml, reintubation, acute respiratory distress syndrome/acute lung injury), neurological (stroke, transient ischemic attack), gastrointestinal (ileus, gastric ulcer, gastrointestinal bleeding, hepatopathy, acute pancreatitis, need of parenteral nutrition), renal (acute kidney injury defined by RIFLE criteria - stage Injury and above) infections defined by clinical picture and the need of systemic antibiotic therapy Scoring systems (Euroscore, TISS 28, APACHE II, SAPS3)

Secondary outcomes:

in-hospital mortality, ICU time further development of MPC algorithm

TIME SCHEDULE:

Year 1- starting the project, establishment of a database, recruitment of patients (800) and processing of partial results Year 2- project review, recruitment of patients (800) and processing of partial results and their presentation Year 3- project review, recruitment of patients (800), final results processing and their publication, study ending

METHODS:

Type of the study: prospective, randomized, controlled, double blinded Inclusion criteria: patients undergoing cardiac surgery, men and women aged 18-90 years, signed informed consent Exclusion criteria: patient's dissent, allergy to insulin or other components added to insulin solution Reasons for exclusion during study: repeated (twice) major hypoglycemia Randomization: on admission to OR into two equally large groups (A, B), after signed informed consent

A = Group of intensive glycemia control: blood glucose level will be maintained by continuous insulin infusion (Actrapid, Novo Nordisk A/S, Bagsvaerd, Danemark - 50 IU/50 ml FR) according to actual glycemia to keep it within normoglycemia limits (4.4 - 6.1 mmol/l) since patient's admission to operating room. Samplings will be taken in 1 to 4 hours intervals in accordance with glycemia stability and MPC algorithm suggestions.

B = Group of standard glycemia control: blood glucose level will be maintained by continuous insulin infusion (see above) within normoglycemia limits (4.4 - 6.1 mmol/l) after patient's admission to ICU after cardiac surgery. During surgery hyperglycemia will not be interfered before it will reach level of 10 mmol/l, then i.v. bolus of 1-2 IU of rapid-acting insulin was administered in order to keep glucose values under this threshold.

Data collection: demographic and clinical characteristics, BMI, standard laboratory findings, perioperative organ complications (respiratory, renal, hematologic, immunologic, infection, wound healing), weaning from ventilatory support, use of catecholamine, in-hospital mortality, scoring (Euroscore, TISS 28, APACHE II, SAPS)

CONCLUSION:

The answer the question when is the optimal time to start glycemia control in patients with in advance known beginning of acute stress reaction would give us a chance, if our hypothesis will be confirmed, to block on time negative effects of hyperglycemia and thereby to decrease number of postoperative organ complications, what would have a significant importance not only medical, but also socio-economical.

Also further eMPC improvement based on clinical data from this study will give to intensivists instrument for markedly simpler and mainly more accurate glycemia normalization and glycemia control in critically ill patients then recent glycemia protocols enable.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery
* men and women
* aged 18-90 years
* signed informed consent

Exclusion Criteria:

* patient's dissent
* allergy to insulin or other components added to insulin solution

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2384 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Morbidity comparison of perioperative vs. postoperative glycemia control | in-hospital
  Number of adverse events from any cause during the postoperative hospital stay

SECONDARY OUTCOMES:
mortality | in-hospital
  in-hospital mortality, ICU time

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blaha, M.D., PhD., Principal Investigator — 1st Faculty of Medicine, Charles University in Prague
Locations (1):
- General University Hospital Prague, Prague, Czechia

REFERENCES:
- [Background] Blaha J, Kopecky P, Matias M, Hovorka R, Kunstyr J, Kotulak T, Lips M, Rubes D, Stritesky M, Lindner J, Semrad M, Haluzik M. Comparison of three protocols for tight glycemic control in cardiac surgery patients. Diabetes Care. 2009 May;32(5):757-61. doi: 10.2337/dc08-1851. Epub 2009 Feb 5. PMID 19196894
- [Background] Hovorka R, Kremen J, Blaha J, Matias M, Anderlova K, Bosanska L, Roubicek T, Wilinska ME, Chassin LJ, Svacina S, Haluzik M. Blood glucose control by a model predictive control algorithm with variable sampling rate versus a routine glucose management protocol in cardiac surgery patients: a randomized controlled trial. J Clin Endocrinol Metab. 2007 Aug;92(8):2960-4. doi: 10.1210/jc.2007-0434. Epub 2007 Jun 5. PMID 17550955
- [Background] Plank J, Blaha J, Cordingley J, Wilinska ME, Chassin LJ, Morgan C, Squire S, Haluzik M, Kremen J, Svacina S, Toller W, Plasnik A, Ellmerer M, Hovorka R, Pieber TR. Multicentric, randomized, controlled trial to evaluate blood glucose control by the model predictive control algorithm versus routine glucose management protocols in intensive care unit patients. Diabetes Care. 2006 Feb;29(2):271-6. doi: 10.2337/diacare.29.02.06.dc05-1689. PMID 16443872
- [Derived] Blaha J, Mraz M, Kopecky P, Stritesky M, Lips M, Matias M, Kunstyr J, Porizka M, Kotulak T, Kolnikova I, Simanovska B, Zakharchenko M, Rulisek J, Sachl R, Anyz J, Novak D, Lindner J, Hovorka R, Svacina S, Haluzik M. Perioperative Tight Glucose Control Reduces Postoperative Adverse Events in Nondiabetic Cardiac Surgery Patients. J Clin Endocrinol Metab. 2015 Aug;100(8):3081-9. doi: 10.1210/jc.2015-1959. Epub 2015 Jun 16. PMID 26079777